CLINICAL TRIAL: NCT05556187
Title: Automated Oxygen Titration in Daily Life of Patients With Chronic Obstructive Pulmonary Disease on Home Oxygen Treatment
Brief Title: Automated Oxygen Titration at Home in Patients With COPD on Home Oxygen
Acronym: DaiLiHOT_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Linette Marie Kofod, Physiotherapist, Primary investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DaiLiHOT_2
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-11

CONDITIONS: COPD; Hypoxemia
Keywords: long term oxygen treatment; Automated oxygen titration; Physiotherapy; Activities of daily living
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a multicentre pilot randomized crossover feasibility trial.
Masking Description: The two different oxygen doses at home is randomised after the initial assessment. It is not possible to blind the patients nor the investigator in this feasibility design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual fixed oxygen dose (No Intervention): * The oxygen dose will be as usual.
  * The patient's activity level will be monitored using SENS.
  * The patient will be asked to wear a wrist pulse oximeter to monitor pulse rate and saturation.
- Automated oxygen titration (Experimental): * The O2matic equipment will be installed in the home of the patients. The SpO2-target will be set at 90-94%
  * The patient's activity level will be monitored using SENS.
  * The patient will be asked to wear a wrist pulse oximeter to monitor pulse rate and saturation and send the information to O2matic. O2matic will adjust the oxygen flow between 0.5-8 l/min according to the algorithm in the devise aiming at the SpO2-target interval.
  * The patients will use their usual portable oxygen devises for use when being active outdoor. They are allowed a higher oxygenflow if needed.
  Interventions: Other: Individualized automated oxygen titration

INTERVENTIONS:
Other: Individualized automated oxygen titration — Automated oxygen titration based on the oxygen saturation during the entire day.
  Arms: Automated oxygen titration

SUMMARY:
Twelwe patients with COPD and long term oxygen treatment (LTOT) will be included in the study. An automated home oxygen titrations (HOT) device will be attached to the patient´s home oxygen equipment. For 2x4 consequent days, the patients will be monitored and saturations, oxygen flow and physical activity level will be registered. In randomized order, the patients will use their usual fixed oxygen dose or automated oxygen titration during the first four days and then crossover. The monitoring consists of a wrist pulse oximeter (register pulse and saturation which is send to the HOT device) and a physical activity sensor attached to the patient's knee. At study start and after both of the four days the patients´dyspnea and QoL will be assessed.

After the study period the patients will in an explorative design based on qualitative methodology be interviewed in order to explore the patients experiences with automated oxygen titration during daily activity and on dyspnea.

DETAILED DESCRIPTION:
Twelve patients with COPD and long term oxygen treatment (LTOT) will be included in the study. The purpose is to evaluate the feasibility of automated oxygen titration during daily living incl. activities. The pilot feasibility design has been chosen as this will be

* the first study testing automated oxygen titration in the patients' home,
* the first study testing automated oxygen titration adjusted not only at rest but during the entire day with the possibility to deliver up to 8 l/min.

Demographic data, will be registered. Oxygen consumption and oxygen saturation (SpO2) will be registered. O2matic Home Oxygen Treatment (HOT) is a device, which based on continuous, non-invasive measurement of SpO2 adjusts oxygen flow to the patient within a defined target interval. SpO2-target can be set individually, but in this study will be fixed at 90 to 94 % with a flow from 0.5-8 l/min. If SpO2 falls below 90 % oxygen flow will increase, and if SpO2 increases above 94 % oxygen flow will decrease. The adjustments are done every second based on average SpO2 for the last 15 seconds.

Blood gas analysis (ABG): Two venous blood sample will be taken, the first with the usual oxygen dose and the second after 20 minutes with an oxygen flow of 8 l/min. The analysis will look at pH-value and the PvCO2.

Clinical COPD Questionnaire (CCQ): 24-hour CCQ measures health status and can be used to assess health-related quality of life (HRQL). It measures symptoms within the last 24 hours as well as functional and mental state, and it is a predictor of mortality in patients with COPD. It is a short questionnaire with 10 items rated on a scale with 6 grades. The items are dyspnea at rest and on exercise, fear of worsening in the condition, depression, cough and sputum, limitations with strenuous and moderate physical activity, limitations with daily activities and social activities. Besides the total score ranging from 0 to 6 there are 3 subscores representing symptoms, mental state and functional state. An improvement of 0.4 is considered clinically significant. CCQ is validated in several languages including danish, and has proven to have good reliability and validity and to be responsive to changes and interventions, such as exacerbations, pulmonary rehabilitation and smoking cessation.

Physical Activity Level: The physical activity will be monitored using A SENS motion® sensor. With a patch above the knee, SENS registers time at rest, standing, walking, steps taken and motion intensity. 600 steps per day has been suggested to be a clinically relevant difference for patients with COPD.

Intervention An O2matic HOT device will be attached to the patient´s home oxygen equipment. For 2x4 consequent days, the patients will be monitored and saturations, oxygen flow and physical activity level will be registered. In randomized order, the patients will use their usual fixed oxygen dose or automated oxygen titration during the first four days and then crossover. The monitoring consists of a wrist pulse oximeter (register pulse and saturation) and a physical activity sensor attached to the patient's knee. At study start and after both of the four days the patients will be assessed using the CCQ.

Baseline visit

1. The patients will be asked to meet for a baseline testing at the hospital. Besides gathering information, two venous blood gases will be taken. The first with the usual oxygen dose and the next after 20 minutes of 8 l/min. The blood sample will be analyzed in order to avoid respiratory acidosis at home (the patients will be excluded if the develop hypercapnia according the exclusion criteria).
2. The randomization will be performed, and the SENS monitor will be attached above the knee.
3. An appointment will be made for a home visit depending on the order of the randomization. The home visits will be made by the primary investigator
4. The patients will be followed for 2x4 days. Four days with usual fixed oxygen dose and four days with automated oxygen titration.

In a "non- pilot" design CCQ could be a primary outcome, which would require 42 patients to show a MCID of 0.4 with a standard deviation = 0.9. A convenience sample of 12 patients is chosen in the present study, as we consider 12 patients to give a clear impression on the use of HOT at home and also a high enough number of patients to gather data on differences on SpO2 interval, CCQ and the activities performed by the patients, well knowing that we cannot expect to detect a difference with high probability.

Continuous variables are examined for normality and analyzed with either paired t-test (in case of normality) or Wilcoxon-signed-rank test (in case of non-normality). IBM SPSS Statistics for Windows, ver. 25.0 will be used for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Verified history of COPD with FEV1/FVC < 0.70 and FEV1 < 50 %
* Hypoxemic at rest (SpO2≤ 90 %) and fulfilment of general national criteria for LTOT

  * Partial pressure of Oxygen (PaO2) (without oxygen supplement) ≤7.3 kPa in clinically stable and optimally treated condition
  * Increase in PaO2 after oxygen supplementation (to 8.0-9.0 kPa) without decrease in arterial pH (> 0.03 kPa)
  * The oxygen is used at least 15 hours daily (optimally 24 hours daily)
  * The treatment is handled by hospital departments with lung medical expertise.
* Able to walk at least 30 meters
* Age >18, Cognitively able to participate in the study and willing to give informed consent

Exclusion Criteria:

* Pulmonary or cardiac condition other than COPD limiting physical performance
* Unstable heart condition or stenotic aortic valve disease
* A physical condition including paralysis, lower extremity pain, or back problem limiting physical performance
* Exacerbation in COPD treated with either antibiotics or prednisolone within the last 3 weeks
* The patients will also be excluded if they have a drop in pH to < 7,31 (venous blood gas) on 8 litres per minute of oxygen flow OR an increase in PvCO2 on > 1 kPa compared to usual fixed oxygen dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of using automated oxygen titration at home | Immediately after the 2x4 days intervention
  Automated oxygen titration during daily living will be considered feasible if
  1. Data is successfully transmitted from the wrist pulse oximeter to O2matic HOT and further to the cloud solution (<10 % data loss).
  2. The patients are wearing the wrist pulse oximeter for more than 50 % of the daytime (08:00 - 20:00)
  3. The time spent within acceptable SpO2-interval is statistically different between arms and in favor of automated oxygen titration with a difference of at least 10 percentage difference in time.
  4. The patients are at least as active with O2matic HOT as with conventional oxygen therapy, measured by SENS activity monitor.
  5. The patients are safe with no serious adverse events, including hypercapnia leading to unscheduled healthcare contacts.

SECONDARY OUTCOMES:
Change in CCQ-score | Immediately after the intervention
  The difference in CCQ-score after four days using automated oxygen titration compared to usual fixed dose.
Physical activity | Immediately after the intervention
  Difference in physical activity level (time spend walking and standing vs sitting or lying). Steps taken.

CONTACTS AND LOCATIONS:
Overall Officials: Linette M Kofod, PT, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Linette Marie Kofod, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
Data access in Denmark are under very strict juristic data protection law. Any possible access or sharing demands a part application to; (1) Danish Data Protection Agency, (2) Ethics Committee of the Capital Region, (3) National Health Data Authorities.
  Only if the applications are approved data will be considered available for sharing.
  The authors will not be able to support this process.